CLINICAL TRIAL: NCT03535129
Title: Investigating a Response Modulation Hypothesis of Socioemotional Processing Associated With Alcohol Use Disorder
Brief Title: A Response Modulation Hypothesis of Socioemotional Processing Associated With Alcohol Use Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 180098; 18-AA-0098
Record Dates: First submitted 2018-05-23; First posted 2018-05-24 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-06-02

CONDITIONS: Healthy Volunteers; Alcohol Drinking Related Problems; Alcohol-Related Disorders
Keywords: Alcohol; Socioemotional; Functional Magnetic Resonance Imaging (fMRI); Neurofeedback; Drug Relapse
MeSH Terms: conditions — Alcohol-Related Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stage 1 (No Intervention): Pilot portion to optimize intervention and achievecorrelational research aims
- Stage 2 (Experimental): Main Clinical Trial with random assignment
  Interventions: Behavioral: Real time fMRI neurofeedback

INTERVENTIONS:
Behavioral: Real time fMRI neurofeedback — During fMRI study, display feedback of brain activity to practice and reinforce control of alcohol craving.
  Arms: Stage 2

SUMMARY:
Background:

Problem drinking affects nearly half the people who drink alcohol. Drinking alcohol affects a person s social behavior and brain structure, but researchers don t have a good understanding of how. They want to test a technique called neurofeedback to learn more about how to treat problem drinking.

Objectives:

To study what happens in the brains of people who drink alcohol when they look at pictures of social things and of alcohol. To learn if people can control brain activity in a magnetic resonance imaging (MRI) scanner and if this helps people with drinking.

Eligibility:

Adults ages 21 65 who have an alcohol use disorder.

Healthy volunteers ages 21 65

Design:

Participants will be screened with

Physical exam

Medical history

Blood, urine, and heart tests

Mental health interview

Questions about their alcohol drinking.

At each session, participants will have:

A urine test for drugs and pregnancy. If they test positive, they cannot participate.

A breath alcohol test and assessment for alcohol withdrawal.

Participants will complete surveys, talk to researchers about behaviors, and play games.

Participants will have MRI brain scans. The scanner is a metal cylinder in a strong magnetic field. They will lie on a table that slides in and out of the scanner for 1 2 hours.

Participants will do tasks in the scanner:

They will look at pictures, sometimes of alcohol.

They will try to hit a goal. Some participants will get feedback during this task. They will see how their brain activity changes or how someone else s changes.

Participants may have follow-up phone questions at least 3 times over about 6 months.

DETAILED DESCRIPTION:
Study Description:

In the first stage, participants will undergo functional magnetic resonance imaging while looking at socioemotional stimuli and alcohol cues and will pilot a neurofeedback training protocol. Personality traits and executive function will also be investigated. In the second stage, inpatient participants with alcohol use disorder will be randomly assigned to receive active or sham neurofeedback. Participants will undergo two functional magnetic resonance imaging sessions including looking at socioemotional stimuli and alcohol cues, resting state fMRI, and real time neurofeedback during alcohol craving. Ability to inhibit attention to alcohol cues and craving will be assessed prior to and following the neurofeedback as well. Participants will be contacted approximately 1 month, 3 months, and 6 months post release from inpatient treatment to assess outcomes.

Objectives:

The purpose of this protocol is to understand the mechanism whereby neural processes of socioemotional cognition associated with alcohol use disorders lead to negative drinking consequences. This study is a two-stage procedure to both provide evidence of a response modulation deficit associated with socioemotional processing in individuals with alcohol use disorder and investigate how moderating that deficit affects socioemotional processing and negative drinking consequences.

Endpoints:

Brain engagement during exposure to socioemotional stimuli, alcohol cues, and neurofeedback training (fMRI-Scan Portion)

ELIGIBILITY:
* INCLUSION AND EXCLUSION CRITERIA:

Stage 1:

INCLUSION CRITERIA:

1. 21 to 65 years old
2. Healthy volunteers only: Consuming on average 7 or less standard drinks/week if female; 14 or less standard drinks/week if male (as determined by the most recent measurement within the past 90 days Alcohol Timeline Followback)
3. AUD participants only: Diagnosed with current moderate to severe alcohol use disorder according to most recent SCID 5 diagnosis

EXCLUSION CRITERIA:

1. Significant history of head trauma or cranial surgery
2. History of neurological disease based on self-report and neuromotor physical exam, conducted by a health care provider, that would interfere with neuroimaging research. Posthoc, clinical MRI scans done according to NIH Clinical Center policy may be reviewed and if there is evidence from that scan of past or current neuroabnormalities that, in the PI or MAI s expert opinion, interfere with research neuroimaging data, the subject may be excluded from data analysis.
3. Physical health concern that would significantly impair or increase the risk of study participation.
4. Healthy volunteers only: Have fulfilled DSM-5 criteria for a current substance or alcohol use disorder
5. Female participants only: Currently pregnant
6. Presence of any ferromagnetic objects in the body that may be aversively affected by or contraindicated for MRI as determined by the NIAAA MRI Safety Screening Questionnaire
7. Any flag on the NIAAA MRI Safety Screening Questionnaire, unless cleared by medically responsible staff (MD/NP)
8. History of non-substance related psychosis
9. Lack of experience with alcohol (defined as less than 3 lifetime drinks reported in history and physical or on Lifetime Drinking History)

Stage 2:

INCLUSION CRITERIA:

1. 21 to 65 years old
2. Inpatient currently seeking treatment for alcohol use disorder

EXCLUSION CRITERIA:

1. Significant history of head trauma or cranial surgery,
2. History of neurological disease based on self-report and neuromotor physical exam, conducted by a health care provider, that would interfere with neuroimaging research.
3. Physical health concern that would significantly impair or increase the risk of study participation.
4. Presence of any ferromagnetic objects in the body that may be aversively

   affected by or contraindicated for MRI as determined by the NIAAA MRI Safety Screening Questionnaire
5. Any flag on the NIAAA MRI Safety Screening Questionnaire, unless cleared by medically responsible staff (MD/NP)
6. History of non-substance related psychosis
7. Female participants only: Currently pregnant

Inpatients who have been admitted into the behavioral unit at the Clinical Center for AUD treatment, maybe considered for this study. Upon completion of consenting procedure, any data necessary (but not readily available) to determine eligibility maybe collected under this study. However, to avoid undue discomfort, burden, and inconvenience, this information, if available, can be gathered from routine clinical care or other NIAAA clinical studies and data up to 30 days prior to the consenting date. Participants who do not satisfy any of the above criteria will not participate in the study procedures at the time. They may be re-scheduled for a future date(s) when they fulfill all inclusion/exclusionary criteria.

We will utilize SCID diagnoses (from other studies such as 14-AA-0181) to determine AUD diagnosis and any potential Axis I disorders. However, for inpatients, since the nursing practice is initially focused on patient detoxification and treatment, the SCID diagnoses might not always take place within the first week of the patient admission to the alcohol unit. This could seriously hamper the subject recruitment in the second stage of this study. We will conduct the MR scan of eligible participants (based on the above inclusion/exclusion criterion) according to study timeline regardless of the availability of SCID diagnoses.

Inpatients are admitted based on the clinical opinion of medical staff that the individual has a pattern of alcohol use disorder. We will enroll inpatients with this opinion but the SCID diagnoses will be completed in order to have consistent research data on symptomology and severity, and to use any potential Axis I disorder as a study confound. Additionally, we will collect information on medications being taken by patients currently or within the last month, including dose, schedule, and timeline. This will be used as a covariate in the statistical design to control for variation associated with these medications.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2018-09-20 (Actual); Primary Completion 2025-03-23 (Actual); Study Completion 2025-03-23 (Actual)

PRIMARY OUTCOMES:
Alcohol Craving | Acute, 1, 3, 6 months
  Self-report craving, change in cue reactivity
Alcohol Attention Bias | Acute, 1, 3, 6 months
  Socioemotional Alcohol Attention Task

SECONDARY OUTCOMES:
Alcohol consumption | 1, 3, 6 months
  Measured by alcohol timeline followback
Community functioning | 1, 3, 6 months
  Measured by Drinker Inventory of Consequences, self-reported employment and residential stability
Antisocial behavior | 1, 3, 6 months
  Specifically, self-reported crime and police contacts, and intimate partner aggression

CONTACTS AND LOCATIONS:
Overall Officials: Abdolreza Momenan, Ph.D., Principal Investigator — National Institute on Alcohol Abuse and Alcoholism (NIAAA)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2018-AA-0098.html